Title: Radial Artery Vasodilation Heat Study

NCT: NCT03620383

Date: 8/27/2019

Statistical Analysis plan:

Statistical analysis will be performed using Stata v14.2 (StataCorp LLC, College Station, TX). Categorical variables and numerical values will be reported as frequencies (percentage) and mean  $\pm$  standard deviation, and compared between two groups using the Chi² test and independent samples t-test, respectively. Trends in radial artery CSA will be compared between PaW and control groups using the repeated measure analysis of variance (rANOVA). P value < 0.05 was considered statistically significant in all analyses.